CLINICAL TRIAL: NCT00575393
Title: A Phase I Dose Escalation Study of the PKC Inhibitor, Aurothiomalate (ATM) in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Gold Sodium Thiomalate in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MC0622; MC0622 (Other: Mayo Clinic Cancer Center); 06-003532 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gold Sodium Thiomalate; Gene Expression Profiling; alovudine; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gold sodium thiomalate
Genetic: gene expression analysis
Other: fluorine F 18 fluorothymidine
Other: mass spectrometry
Other: pharmacological study

SUMMARY:
RATIONALE: Gold sodium thiomalate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of gold sodium thiomalate in treating patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose of gold sodium thiomalate in patients with advanced non-small cell lung cancer.
* To describe the toxicities associated with this treatment.
* To describe any preliminary evidence of biologic activity.
* To further assess the correlation between PKCι expression and the antitumor effects of gold sodium thiomalate.
* To study the association of clinical (toxicity and/or tumor response or activity) with pharmacokinetic/pharmacodynamic parameters.
* To describe anti-proliferative activity of gold sodium thiomalate through 3-deoxy-3-[^18F]-fluorothymidine positron emission tomography imaging.

OUTLINE: This is a dose-escalation study of gold sodium thiomalate.

Patients receive gold sodium thiomalate intramuscularly on days 1, 8, 15 and 22. Treatment repeats every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive gold sodium thiomalate once every 4 weeks until a total cumulative dose of 1 gram is delivered.

Blood samples are collected at baseline and prior to therapy in weeks 3, 5, 7, 9, and 11. Samples are analyzed by mass spectometry for pharmacokinetics. Paraffin-embedded tumor tissue samples are analyzed for PKC_l expression and antitumor activity. Antiproliferative effects of gold sodium thiomalate are analyzed by 3-deoxy-3-[^18F]-fluorothymidine positron emission tomography imaging.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced non-small cell lung cancer
* No known standard therapy for disease that is potentially curative or definitely capable of extending life expectancy
* No symptomatic or worsening CNS metastases despite optimal therapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 3 times ULN (5 times ULN if liver involvement)
* Creatinine ≤ 1.2 times ULN
* Hemoglobin ≥ 9.0 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be willing to provide blood and tissue samples
* No uncontrolled infection
* No New York Heart Association class III or IV heart disease
* No known allergy to gold sodium thiomalate

PRIOR CONCURRENT THERAPY:

* Recovered from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* No prior chemotherapy within the past 3 weeks
* No prior mitomycin C or nitrosoureas within the past 6 weeks
* No prior immunotherapy within the past 3 weeks
* No prior biologic therapy within the past 3 weeks
* No prior radiotherapy within the past 3 weeks
* No prior radiotherapy to > 25% of bone marrow
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (i.e., utilized for a non-FDA-approved indication and in the context of a research investigation)
* No concurrent prophylactic colony stimulating factors

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-01-25 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2012-02-14 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Toxicity
Biologic activity
Correlate PKCl expression with antitumor effects of gold sodium thiomalate
Correlate toxicity and/or tumor response or activity with pharmacokinetic and pharmacodynamic parameters
Anti-proliferative activity of gold sodium thiomalate by PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, MD, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota